CLINICAL TRIAL: NCT06519734
Title: Primitive Immunodeficiency, Intrauterine Devices and Menstrual Hygiene Products
Acronym: FEMIDIP
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240435; 2024-A00635-42 (Other: IDRCB Number)
Record Dates: First submitted 2024-07-19; First posted 2024-07-25 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Primary Immune Deficiency Diseases
Keywords: Primary immune deficiency diseases; Contraception; Intrauterine device; Menstrual hygiene products; Menstrual cups; Tampons; Infectious complications
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Adult women registered in the Center for Hereditary Immune Deficits (CEREDIH), hospital Necker-Enfants Malades, Paris.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire intended for patients on contraceptive modalities and use of menstrual hygiene products.
  Consultation of the medical records of patients who have reported infectious complications linked to the use of intrauterine devices, tampons or menstrual cups.

SUMMARY:
Primary immune deficiency diseases (PIDDs) constitute a large group of genetic disorders of the immune system which associates to varying degrees an increased susceptibility to infections and immuno-pathological manifestations: allergy, inflammation, autoimmunity, lymphoproliferation, malignancy.

Although their prevalence remains underestimated, there has been an increase in cases diagnosed in the last 10 years. The national average prevalence is 8.6 patients per 100,000 inhabitants with an incidence of 400 new cases per year in France. Life expectancy varies depending on the type of deficiency, and its impact in terms of infectious complications or malignancy.

With therapeutic progress, life expectancy increases, and more patients are concerned by contraception and menstrual hygiene. Due to the lack of data and for fear of an infectious complication, the use of intrauterine devices (IUD) and tampons or menstrual cups is traditionally advised against in patients with PID.

The objective of the research is to study the contraception methods and menstrual hygiene products used by patients with primary immunodeficiency and to evaluate related infectious complications.

The contraceptive methods of these patients, the occurrence of upper genital infections associated with the use of an intrauterine device, the severity and the evolution of these infections will be evaluated. A possible refusal to insert an intrauterine device by a healthcare professional due to primary immunodeficiency will also be studied.

Likewise, the types of menstrual hygiene products used will be studied - napkins, menstrual cups, tampons, menstrual panties -, as well as the possible occurrence of associated infectious complications - in particular menstrual toxic shock syndrome, and the treatment, severity and evolution of these complications.

DETAILED DESCRIPTION:
Primary immune deficiency diseases (PIDDs) constitute a large group of genetic disorders of the immune system which associate to varying degrees an increased susceptibility to infections and immuno-pathological manifestations: allergy, inflammation, autoimmunity, lymphoproliferation, malignancy.

Although their prevalence remains underestimated, there has been an increase in cases diagnosed in the last 10 years. The national average prevalence is 8.6 patients per 100,000 inhabitants and the incidence is 400 new cases per year in France. Life expectancy varies depending on the type of deficiency, and its impact in terms of infectious complications or malignancy.

With therapeutic progress, life expectancy increases and more patients are concerned by contraception and menstrual hygiene. Due to the lack of data and for fear of an infectious complication, the use of intrauterine devices (IUD) and tampons or menstrual cups is traditionally not recommended in patients with PID.

IUDs are one of the most effective, long-lasting and low-cost methods of contraception, which have the major advantage of causing few drug interactions. Access to effective and appropriate contraception is a major issue for patients with PID because these patients have high-risk pregnancies. Multidisciplinary pregnancy planning allows for adaptation of anti-infective treatments and prophylaxis. These patients often have medication that may interfere with oral contraception, so IUDs could provide many benefits. The incidence of upper genital infections after insertion of an IUD in the general population is 1.6 cases per 1000 patient-years, with a risk 6 times higher in the 20 days after insertion. The risk of developing an upper genital infection is linked to the breakdown of the cervical mucus barrier and the introduction of bacteria from the lower genital tract into the uterine cavity.

The main infectious complication associated with the use of intravaginal menstrual protection is menstrual toxic shock syndrome, a rare but serious pathology caused by the production of the TSST-1 toxin by Staphylococcus aureus. The use of a tampon is one of the main risk factors identified and menstrual cups do not seem to be less likely to promote menstrual toxic shock syndrome. These risks lead to the use of tampons and menstrual cups being discouraged in patients with PID. However, there are no data in the literature on the association between immunosuppression and increased risk of menstrual toxic shock syndrome. Additionally, adult patients with PID will likely use these menstrual hygiene products during their lifetime.

It is therefore crucial to better characterize the risks incurred by patients with PID and the potential infectious complications associated with these devices.

The objective of the research is to study the contraception methods and menstrual hygiene products used by patients with primary immunodeficiency and to evaluate related infectious complications.

The contraceptive methods of these patients, the occurrence of upper genital infections associated with the use of an intrauterine device, the severity and the evolution of these infections will be evaluated. A possible refusal to insert an intrauterine device by a healthcare professional due to primary immunodeficiency will also be studied.

Likewise, the types of menstrual hygiene products used will be studied - napkins, menstrual cups, tampons, menstrual panties -, as well as the possible occurrence of associated infectious complications - in particular menstrual toxic shock, and the treatment, the severity and the evolution of these complications.

ELIGIBILITY:
Inclusion Criteria:

* Adult woman with primary immune deficiency disease and registered in the reference Center for Hereditary Immune Deficits (CEREDIH, hospital Necker-Enfants Malades, Paris)
* Patient not opposed to participation in research

Exclusion Criteria:

* Refusal to participate of the study
* Deceased patient
* Minor patient
* Patient under legal protection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Female patients with primary immune deficiency disease included in the CEREDIH (reference Center for Hereditary Immune Deficits) national cohort.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Occurrence of infectious complications associated with the use of intrauterine devices and tampons or menstrual cups in patients with primary immunodeficiency | Time 0
  Occurrence of an infectious complication - upper genital infection or menstrual toxic shock - associated with the use of an intrauterine device, tampon or menstrual cup in patients with primary immunodeficiency.
  These complications will be declared by patients via the study questionnaire and then confirmed by consultation of the medical file.

SECONDARY OUTCOMES:
Frequency of use of intrauterine devices, menstrual cups and tampons in patients with primary immunodeficiency | Time 0
  Frequency of use of intrauterine devices, menstrual cups or tampons reported by patients on the study questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Charlier-Woerther, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Aude Beloeuvre, MD, Study Director — Assistance Publique - Hôpitaux de Paris; Nizar Mahlaoui, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No